CLINICAL TRIAL: NCT02381106
Title: The ADRB3 Adrenergic Receptor - a Possible New Target for Controlling Pre-eclampsia and Hypertension in Pregnancy and Uterine Contractions in Non-pregnant and Pregnant Myometrium
Brief Title: The ADRB3 Receptor in Pregnancy
Status: Suspended | Type: Observational
Why Stopped: assay difficulties
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Helena Kopp Kallner, MD, PhD, Karolinska Institutet
Other Study IDs: VAI
Record Dates: First submitted 2014-11-11; First posted 2015-03-06 (Estimated); Last update posted 2023-05-17 (Actual); Status verified 2023-05

CONDITIONS: Pregnancy Complications
Keywords: arterial contractility; Uterine contractility
MeSH Terms: conditions — Pregnancy Complications

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — uterine specimen placental specimen
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Women with preeclampsia: Women delivered by cesarian section and with preeclampsia
- Women with dysfunctional labor: Women delivered with cesarian section due to dtsfunctional labor
- Women with cesarian section due to maternal request: Women with cesarian section due to maternal request
- Women with preamture labor: Women with pemature labor undergoing cesarian section

SUMMARY:
The primary overall objective of this study is to characterize the levels of and compare levels of the ADRB3 receptor in human non-pregnant myometrium, pregnant myometrium at different time points in pregnancy, in normal and dysfunctional labor and also to measure levels and expression of these receptors in placental arteries at different maturation statuses of placenta and in pre-eclampsia/hypertension

ELIGIBILITY:
Inclusion Criteria:

* Women undergoing cesarian section

Exclusion Criteria:

* Interkurrent diseases

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Pregant women undergoing cesarian section.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2014-11; Primary Completion 2028-12 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
characterization of the levels of the ADRB3 receptor in human pregnant myometrium | 1 month

CONTACTS AND LOCATIONS:
Locations (1):
- Dept of Obstetrics and Gynecology, Danderyd Hospital, Stockholm, Sweden